CLINICAL TRIAL: NCT06456229
Title: Time to Return of Bowel Function Following Perioperative Probiotics in Colorectal Cancer Surgery (PICCS-1)
Brief Title: Time to Return of Bowel Function Following Perioperative Probiotics in Colorectal Cancer Surgery
Acronym: PICCS-1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024/00180
Record Dates: First submitted 2024-06-06; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Colorectal Cancer; Ileus Postoperative; Flatus; Diet, Healthy
Keywords: colorectal cancer; colorectal surgery; nutritional supplementation; probiotics; time to bowel movement; time to flatus; length of stay; complications
MeSH Terms: conditions — Colorectal Neoplasms; Flatulence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (No Intervention): Control arm with no nutritional supplementation
- Arm 2 (Active Comparator): Control arm with nutritional supplementation but without probiotics
  Interventions: Dietary Supplement: Nestle Isocal
- Arm 3 (Experimental): Nutritional supplementation with probiotics
  Interventions: Dietary Supplement: Nestle Boost Optimum

INTERVENTIONS:
Dietary Supplement: Nestle Isocal — Nestle Isocal
  Arms: Arm 2
Dietary Supplement: Nestle Boost Optimum — Nestle Boost Optimum
  Arms: Arm 3

SUMMARY:
There is pre-existing evidence that probiotics could be useful in the improvement of ileus rates. One metaanalysis of 30 studies demonstrated a reduction in the prevalence of post-operative ileus as determined by time to flatus, time to defecation, as well as postoperative abdominal distension (PMID:37373843). More broadly in gastrointestinal surgery, a meta-analysis of 21 randomised controlled trials similarly affirmed the speedier recovery of gastrointestinal function after surgery when probiotics were administered (PMID: 35231076). In spite of these advantages, the routine use of probiotics perioperatively for colorectal cancer surgery is not performed in Singapore. We therefore seek to perform a trial to investigate whether probiotic administration perioperatively may reduce post operative ileus rates.

ELIGIBILITY:
Inclusion Criteria:

1. undergoing elective colorectal cancer surgery in which an oncologic resection is planned
2. age between 21 and 99 years at the time of consent
3. willing to consider oral nutritional supplementation
4. on an early recovery after surgery (ERAS) pathway
5. able to provide informed consent

Exclusion Criteria:

1. patients with known contraindications to probiotic use
2. patients undergoing emergency surgery
3. taking any other form of probiotics
4. taking oral antibiotics within 7 days of commencement of study
5. vulnerable patients including pregnant patients, inmates, and those who are cognitively impaired and therefore are not able to provide informed consent.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Time to bowel movement | 0 - 14 days
  This records the number of days from the day of surgery before the first bowel movement was experienced by the patient.

SECONDARY OUTCOMES:
Time to flatus | 0 - 14 days
  This records the number of days from the day of surgery before the first flatus was experienced by the patient.
Adverse events | From commencement of the intervention to 30 days after surgery
  Any adverse events related to the intervention. This comprises predominantly gastrointestinal related complications
Infective complications | From date of surgery to 30 days after surgery
  Any infective complications which may occur in the postoperative period.
Length of hospital stay | 0 - 14 days
  This records the number of days following surgery before the patient is discharged.

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.

REFERENCES:
- [Derived] Chan DKH, Siew BE, Lau J, Koh J, Lee MX, Ang C, Pang NQ, Tan KK. Time to return of bowel function following perioperative probiotics in colorectal cancer surgery (PICCS-1): study protocol for a randomized controlled trial. Trials. 2025 Feb 19;26(1):60. doi: 10.1186/s13063-025-08773-2. PMID 39972354